CLINICAL TRIAL: NCT03064451
Title: Repetitive Activation Patterns and Focal Impulses Identification and Ablation in Persistent AF Using the RHYTHMFINDER-192
Brief Title: Repetitive Activation Patterns and Focal Impulses Identification and Ablation in Persistent AF
Acronym: RAPID-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPID-AF
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation - ablation procedure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): cartofinder guided ablation followed by PVI
  Interventions: Procedure: cartofinder guided ablation followed by PVI

INTERVENTIONS:
Procedure: cartofinder guided ablation followed by PVI — cartofinder guided ablation followed by PVI

SUMMARY:
The primary purpose of this study is to assess the effectiveness of using CARTOFINDER™ maps created by the RHYTHMFINDER-192 catheter and the CARTOFINDER™ Algorithm to terminate persistent atrial fibrillation (PsAF) to either Normal Sinus Rhythm or Atrial Tachycardia compared to pulmonary vein isolation (PVI) in treating PsAF. The RHYTHMFINDER-192 catheter is investigational, while the CARTOFINDER™ system is CE marked in Europe.

All subjects with persistent AF who are scheduled to undergo a clinically indicated ablation procedure for management of their persistent AF will be the target population for screening. The study will enroll approximately 40-70 subjects. Subjects will undergo CARTOFINDER™ guided ablation (CFGA) followed by PVI. Subjects will have follow-up visits at 7 days, 3, 6 and 12 months postprocedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Patients who have signed the Patient Informed Consent Form (ICF)
3. Scheduled to undergo a clinically-indicated catheter ablation procedure for treatment of

   1. persistent atrial fibrillation (defined as continuous atrial fibrillation that is sustained beyond seven consecutive days).
   2. drug-resistant atrial fibrillation. (failed 1 or more class I or III antiarrhythmic drugs) and demonstrating Persistent AF (requiring drugs or electrical shock to terminate AF)
4. In AF at the time of the baseline CARTOFINDER™ Map (spontaneous)
5. Left Atrium (LA) must demonstrate sufficient electrical activity to allow for the identification of ablation targets.
6. Able and willing to comply with all pre-, post-, and follow-up testing and requirements (e.g. patients not confined by a court ruling)

Exclusion Criteria:

1. Paroxysmal Atrial Fibrillation
2. Continuous AF > 12 months (1-Year) (Longstanding Persistent AF) Subjects previously diagnosed as Long Standing Persistent (LSP) but have demonstrated the ability to maintain Normal Sinus Rhythm for >30 days after cardioversion and have not been in AF greater than 1 year at the time of the procedure remain eligible for inclusion.
3. Previous ablation procedure for PsAF (defined as ablations involving more than only PV isolation)
4. Patients with a left atrial size >55 mm (echocardiography, parasternal long axis view).
5. Inability to restore sinus rhythm for 30 seconds or longer in the opinion of the investigator.
6. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
7. Atrial arrhythmia patients with structural atrial disease such as a prior history of atriotomy from prior atrial surgery, presence of an atrial septal defect, and/or presence of an atrial septal closure patch.
8. History of or current blood clotting or bleeding abnormalities, contraindication to systemic anticoagulation (i.e., heparin, warfarin, dabigatran, or a direct thrombin inhibitor).
9. significant pulmonary disease, cardiac surgeries, unstable angina, uncontrolled heart failure, acute illness or systemic infection, or any other disease or malfunction that would preclude treatment in the opinion of the investigator.
10. Current enrollment in a study evaluating another device or drug.
11. A complex arrhythmia secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
12. Any cardiac surgery within the past 60 days (2 months) (includes PCI)
13. Subjects that have ever undergone valvular cardiac surgical procedure (i.e., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
14. Prior ICD or pacemaker implanted
15. Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation.
16. Presence of a condition that precludes vascular access.
17. Subject has a contra-indication to the device under study per the IFU
18. Women of child bearing potential whom are pregnant, lactating, or planning to become pregnant during the course of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Belgium (3):
  - OLV Aalst, Aalst
  - AZ Sint-Jan Brugge, Bruges
  - Universitair Ziekenhuis Antwerpen, Edegem
- Southlake Regional Health Centre, Newmarket, Ontario, Canada
- Nemocnice České Budějovice, České Budějovice, Czechia
- United Kingdom (2):
  - St Bartholomew's hospital, London
  - London Health Sciences Center, London

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Persistent Atrial Fibrillation (PsAF): Participants with PsAF and an ablation target on the CARTOFINDER (CF) map underwent CARTOFINDER-Guided Ablation (CFGA) followed by Pulmonary Vein Isolation (PVI) Wide Area Circumferential Ablation (WACA) ablation and followed-up at 7 days, 3 months, 6 months, and 12 months post ablation procedure. Participants not displaying an ablation target on CARTOFINDER were treated per investigator's standard of care and followed up until 7 days post-procedure.
Period: Overall Study
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Started | 60
Safety Population | 52
Completed | 46
Not Completed | 14
Not completed — Lost to Follow-up | 1
Not completed — Mapping Failure | 4
Not completed — Exited prior to procedure | 8
Not completed — Withdrew consent: 3-month FU visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Acute Success Post CartoFinder Guided Ablation (CFGA) Only (Before Pulmonary Vein Isolation [PVI] and Without Cardioversion).
Description: Acute success defined as rate of conversion of Atrial Fibrillation to Normal Sinus Rhythm or Atrial Tachycardia, after CARTOFINDER Guided Ablation (CFGA) only (before Pulmonary Vein Isolation [PVI] and without cardioversion).
Time Frame: Up to 7 days
Population: The evaluable participant population included all enrolled participants who had the RHYTHMFINDER 192 Catheter inserted and where CARTOFINDER-guided ablation was performed.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 48
Percentage of participants | 22.9

2. Primary Outcome: Percentage of Participants With Acute Success Post CartoFinder Guided Ablation (CFGA) and Pulmonary Vein Isolation (PVI) Without Cardioversion
Description: Acute success defined as rate of conversion of Atrial Fibrillation to Normal Sinus Rhythm or Atrial Tachycardia, after CFGA and PVI without Cardioversion.
Time Frame: Up to 7 days
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 48
Percentage of participants | 33.3

3. Primary Outcome: Percentage of Participants With Procedural Success
Description: Procedural success defined as the conversion of Atrial Fibrillation to Normal Sinus Rhythm or Atrial Tachycardia after overall ablation procedure, with or without the need for cardioversion.
Time Frame: Up to 7 days
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 48
Percentage of participants | 97.9

4. Primary Outcome: Percentage of Participants With Recurrence of Atrial Fibrillation, Atrial Flutter, and Atrial Tachycardia Episodes of Greater Than or Equal to (>=) 30 Seconds to Measure the Effectiveness Success Rate for up to 12 Months
Description: Documented AF/AT/AFL recurrence is defined as any occurrence of documented (symptomatic) atrial fibrillation, atrial flutter, and atrial tachycardia episodes >= 30 seconds during the post-blanking period (Day 91-365). Here 'HM' signifies Holter monitoring.
Time Frame: Up to 12 months
Population: Evaluable population:enrolled participants who had RHYTHMFINDER 192 Catheter inserted, where CFGA performed. 'N' (Number of participants analyzed):number of participants who completed 12 months follow-up(post initial ablation) or data collected from ElectroCardioGram, HM, or Post Procedure Arrhythmia Log forms beyond 337 days post index procedure.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 47
Percentage of participants | 72.3

5. Primary Outcome: Number of Participants With Early-onset Primary Adverse Events
Description: Incidence of early-onset (within 7 days of the initial mapping and ablation procedure) Primary Adverse Events (PAEs) was reported. PAEs included death, Atria-Esophageal Fistula, Cardiac Tamponade/Perforation, Myocardial Infarction, Stroke/Cerebrovascular Accident, Thromboembolism, Transient Ischemic Attack, Diaphragmatic Paralysis, Pneumothorax, Heart Block, Pulmonary Vein Stenosis, Pulmonary Edema (Respiratory Insufficiency), Pericarditis and Major Vascular Access Complication/Bleeding.
Time Frame: Up to 7 days
Population: The safety participants population included all enrolled participants who had the RHYTHMFINDER 192 Catheter inserted, regardless if CARTOFINDER-guided ablation was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 52
Participants
  Cardiac tamponade / Perforation | 2
  Major vascular access complications / bleeding | 2
  Pericarditis | 1
  Atrio-Esophageal Fistula | 0
  Death | 0
  Diaphragmatic Paralysis | 0
  Heart Block | 0
  Myocardial Infarction | 0
  Pneumothorax | 0
  Pulmonary Edema (Respiratory Insufficiency) | 0
  Pulmonary Vein Stenosis | 0
  Stroke / Cerebrovascular Accident | 0
  Thromboembolism | 0
  Transient Ischemic Attack | 0

6. Secondary Outcome: Number of Participants With Confirmed Entrance Block After Adenosine/Isoproterenol Challenge
Description: Number of participants with confirmed entrance block after adenosine/isoproterenol challenge was reported.
Time Frame: Up to 12 months
Population: Evaluable participant population included all enrolled participants who had the RHYTHMFINDER 192 Catheter inserted and where CARTOFINDER-guided ablation was performed. Here 'N' number of participants analyzed included participants with adenosine/isoproterenol challenge and non-missing confirmation of entry block data collected from the PVI form.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 16
Participants | 15

7. Secondary Outcome: Change of Intra-cycle Length From Pre-CFGA (Baseline) to Post-CFGA and Post-PVI
Description: Change of intra-cycle length from pre-CFGA to post-CFGA and post-PVI is reported to measure the slowing for the overall Atrial Fibrillation rate in both atrium's.
Time Frame: Pre-CFGA (Baseline) to Post-CFGA and Post-PVI (Up to 7 days)
Population: Evaluable participant included all enrolled participants who had RHYTHMFINDER 192 Catheter inserted, where CARTOFINDER-guided ablation was performed. Here 'n' (number analyzed) included participants analyzed at specified categories for post-CFGA and post PVI.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 48
milliseconds
  Left Atrium: Change post-CFGA: number analyzed (Participants) | 41
  Left Atrium: Change post-CFGA | 64.0 (273.62)
  Left Atrium: Change post-PVI: number analyzed (Participants) | 34
  Left Atrium: Change post-PVI | 464.0 (1009.44)
  Right Atrium: Change post-CFGA: number analyzed (Participants) | 26
  Right Atrium: Change post-CFGA | 33.3 (103.58)
  Right Atrium: Change post-PVI: number analyzed (Participants) | 26
  Right Atrium: Change post-PVI | 525.2 (1120.70)

8. Secondary Outcome: Number of Participants With Serious Adverse Device Effects (SADEs) up to 12 Months
Description: Any serious adverse event which was related to the device and/or the procedure was defined as a SADE.
Time Frame: Up to 12 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 52
Participants | 6

9. Secondary Outcome: Number of Participants With All Serious Adverse Events (SAEs) up to 12 Months
Description: Number of participants with SAEs will be evaluated. An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life threatening experience, is a congenital anomaly/birth defect, is suspected transmission of any infectious agent via a medicinal product, is medically important, and may jeopardize participant or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 12 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 52
Participants | 10

10. Secondary Outcome: Number of Participants With Adverse Device Effects (ADEs) up to 12 Months
Description: Number of participants with adverse device effects was reported. Adverse Device Effect (ADE's) are adverse events related to the use of an investigational medical device. This definition includes adverse events resulting from insufficient or inadequate instructions for use deployment, implantation, installation, or operation, or any malfunction of the investigational medical device. This definition includes any event resulting from use errors or from intentional misuse of the investigational medical device.
Time Frame: Up to 12 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 52
Participants | 20

11. Secondary Outcome: Number of Participants With Procedural Related Serious Adverse Event and Non-serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with treatment and therefore can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with use of a medicinal product, whether or not related to that medicinal product. TEAEs were defined as AEs that were reported or worsened on after start of study drug(s) dosing through safety follow-up visit. A serious adverse event (SAE) is any untoward medical occurrence that at any dose resulting in any of following outcomes: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to 12 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
Number analyzed (Participants) | 52
Participants
  Serious Adverse event | 6
  Adverse event | 14

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: The safety participants population included all enrolled participants who had the RHYTHMFINDE 192 Catheter inserted, regardless if CARTOFINDE-guided ablation was performed.
Arm/Group | Participants With Persistent Atrial Fibrillation (PsAF)
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 10/52
Other Adverse Events (participants affected / at risk) | 6/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Persistent Atrial Fibrillation (PsAF) (N=52)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Persistent Atrial Fibrillation (PsAF) (N=52)
Haematoma (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT03064451/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03064451/SAP_001.pdf